CLINICAL TRIAL: NCT05396378
Title: Early Recovery After Cesarean Delivery - Maternal Glucose Homeostasis Following Preoperative Glucose Dose in Diabetic Parturients
Brief Title: Early Recovery After Cesarean Delivery - Maternal Glucose Homeostasis Following Preoperative Glucose Dose
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Women's Hospital HUS (Other)
Responsible Party: Principal Investigator, Antti Vaananen, PRincipal investigator, Women's Hospital HUS
Other Study IDs: Tutkimussuunnitelma_250322_III
Record Dates: First submitted 2022-05-27; First posted 2022-05-31 (Actual); Last update posted 2023-04-25 (Actual); Status verified 2023-04

CONDITIONS: Gestational Diabetes; Cesarean Section Complications
MeSH Terms: conditions — Diabetes, Gestational | interventions — Glucose

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Gestational diabetes: Any parturient who after information agrees to participate in the study. The treatment of the gestational diabetes may be by diet, metformin or insulin according to the hospital's normal protocol.
  Interventions: Dietary Supplement: Oral glucose in liquid form
- Type II diabetes: Any parturient who after information agrees to participate in the study. The treatment of the diabetes may be by diet, metformin or insulin according to the hospital's normal protocol.
  Interventions: Dietary Supplement: Oral glucose in liquid form

INTERVENTIONS:
Dietary Supplement: Oral glucose in liquid form — A glucose containing drink that has a fixed dose of 25 g of glucose per can.
  Other Names: Pre-op drink

SUMMARY:
Diabetic parturients planned for cesarean delivery will be recruited for the study. They will receive a fixed glucose dose to mimize the effects of fasting preoperatively and their blood glucose levels will be monitored.

DETAILED DESCRIPTION:
Informed voluntary parturients planned for cesarean delivery will be informed about the study. The parturients will get prepacked glucose drink containing 100 g and 50 g glucose, respectively. They will consume the 100 g of glucose the night before the planned operation and the 50 g on the morning of the planned cesarean delivery. Their blood glucose level will be monitored by percutaneous continuous blood glucose monitoring every 30 minutes for 2 hours following the glucose dose in the evening and for four hours in the morning of the operation.

The subjective well being of these parturients will be also qualitatively assessed.

ELIGIBILITY:
Inclusion Criteria:

* Volunteers to participate in the study
* Diabetes, either gestational or type II
* Planned for cesarean delivery

Exclusion Criteria:

* Type I diabetes

Ages: 18 Years to 55 Years | Sex: Female
Age Groups: Adult
Study Population: Diabetic parturients excluding type I diabetics who visit the Helsinki University Central Hospital/Women's hospital for the treatment of their diabetes during pregnancy and are planned for cesarean delivery.
Sampling Method: Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2023-07-01 (Estimated); Primary Completion 2023-12-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Increase of blood glucose following the oral glucose dose | 4 hours
  The effect of oral glucose dose on the parturient's blood glucose level (mM)

SECONDARY OUTCOMES:
Maternal subjective well being after oral glucose dose during the preoperative fasting period | 4 hours
  subjective assessment by the parturient (categorial)

CONTACTS AND LOCATIONS:
Locations (1):
- HUS/Women's hospital dept of obstetrics, Helsinki, Finland

IPD SHARING:
Plan to Share IPD: No